CLINICAL TRIAL: NCT06440499
Title: Prenatal Ultrasonographic Screening of Congenital Anomalies of Kidney and Urinary Tract During the Third Trimester of Pregnancy
Brief Title: Screening of Congenital Anomalies of Kidney
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Salah, Assiut University, Assiut University
Other Study IDs: congenital anomalies of kidney
Record Dates: First submitted 2024-05-24; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Kidney Congenital Anomalies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: US — Us

SUMMARY:
To evaluate the role of ultrasound in prenatal diagnosis of congenital anomalies of kidney and urinary system in third trimester of pregnancy.

Primay outcomes:

To determine incidence of congenital anomalies in kidney and urinary system in Third Timerter by ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* • Singleton pregnancy.

  * Healthy women Aged between 20 to 40 years old.
  * Third trimester

Exclusion Criteria:

* • Multiples pregnancies.

  * Maternal D.M or HTN
  * Patients' refusal to participate.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: pregnant
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-03-05 (Estimated); Study Completion 2025-04-05 (Estimated)

PRIMARY OUTCOMES:
To determine sensitivity, spacificy, the +ve PP &-ve P.P of ultrsound screening for renal anomalies. | 1 year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Hamed MH, Sayer JA, Alsahan N, Tulbah M, Kurdi W, Ambusaidi Q, Ali W, Imtiaz F. Novel loss of function variants in FRAS1 AND FREM2 underlie renal agenesis in consanguineous families. J Nephrol. 2021 Jun;34(3):893-900. doi: 10.1007/s40620-020-00795-0. Epub 2020 Jul 8. PMID 32643034